## STATISTICAL ANALYSIS PLAN

## TITLE: Postpartum Non-pharmacologic Pain Management – Randomized Controlled Trial

**INVESTIGATORS:** Sheela Barhan, MD (PI), Rose Maxwell, PhD, Samantha Younglove, DO, Elena Wysong, MD

July 27, 2022

NCT03903172

Statistical analysis will consist of comparison of the study groups (Abdominal binder vs Standard of care) on:

- 1) baseline characteristics including age and baseline pain score.
- 2) study outcomes for average pain score on postpartum day 0 and postpartum day 1.
- 3) postpartum non-narcotic pharmacologic medication use.
- 4) narcotic pharmacologic pain medication used.

Analysis will be as follows:

- 1) Baseline age and postpartum pain scores will be analyzed using Student's T-test.
- 2) Average pain scores on PPD0 and PPD1 will be analyzed using Student's T-test.
- 3) Postpartum non-narcotic pharmacologic medications will be compared using Chi square.
- 4) Post partum narcotic pharmacologic medication use will be analyzed using Fisher's Exact test.